CLINICAL TRIAL: NCT06608732
Title: Clinical Study of Inaticabtagene Autoleucel Combined With Autologous Hematopoietic Stem Cell Transplantation for Adolescents or Adults With MRD-Positive B-Cell Acute Lymphoblastic Leukemia in Initial Complete Remission.
Brief Title: Combination of Inaticabtagene Autoleucel With Autologous Hematopoietic Stem Cell Transplantation for Adolescents or Adults With MRD-Positive B-Cell Acute Lymphoblastic Leukemia in Initial Complete Remission.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024037
Record Dates: First submitted 2024-09-10; First posted 2024-09-23 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Inaticabtagene autoleucel; autologous hematopoietic stem cell transplantation; Minimal Residual Disease
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inaticabtagene autoleucel Combined with Autologous Hematopoietic Stem Cell Transplantation (Experimental)
  Interventions: Biological: Inaticabtagene autoleucel

INTERVENTIONS:
Biological: Inaticabtagene autoleucel — CNCT19 combined with autologous hematopoietic stem cell transplantation，Dose: （0.5 -2）x 10^6/kg CNCT19 Cell Injection via intravenous infusion.

SUMMARY:
Evaluate the safety and efficacy of Inaticabtagene autoleucel combined with autologous hematopoietic stem cell transplantation in adolescents or adults with MRD-positive initial complete remission in B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Evaluate the safety and efficacy of Inaticabtagene autoleucel combined with autologous hematopoietic stem cell transplantation in adolescents or adults with MRD-positive initial complete remission in B-cell acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score of 0 to 1
* Newly diagnosed Ph-negative B-ALL within 6 months, achieving CR1 after standard induction chemotherapy, undergoing at least one consolidation therapy, and patients with bone marrow MRD ≥ 0.01% detected by routine flow cytometry.
* Or newly diagnosed Ph-positive B-ALL within 6 months, achieving CR1 after guideline-recommended induction chemotherapy (or use of TKI), undergoing at least one consolidation therapy, and patients with BCR-ABL1 > 0% detected by routine q-PCR technology.
* No significant organ dysfunction
* Willing and meet the conditions for autologous hematopoietic stem cell transplantation

Exclusion Criteria:

* Burkitt lymphoma/leukemia, heterozygous or double-expressor leukemia, or chronic myeloid leukemia in blast phase.
* Before screening or pre-treatment, bone marrow or peripheral blood with blasts ≥ 5%; or extramedullary leukemia.
* Individuals who have received CAR-T cell therapy before screening or pre-treatment; or patients who have undergone hematopoietic stem cell transplantation.
* Patients with associated genetic syndromes related to bone marrow failure, such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndromes.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival | From autologous hematopoietic stem cell transplantation to 2 years after transplantation
  The time from the start of infusion of Inaticabtagene autoleucel until the diagnosis of relapse or any death (whichever comes first).

SECONDARY OUTCOMES:
Overall survival rate | From autologous hematopoietic stem cell transplantation to 2 years after transplantation
Cumulative recurrence rate | From autologous hematopoietic stem cell transplantation to 2 years after transplantation
MRD negativity rate | 28 days after the first CAR-T cell reinfusion

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No